CLINICAL TRIAL: NCT00813878
Title: Optical Biosensor for the Early Detection of Breast Cancer
Brief Title: Nipple Secretion Samples in Detecting Breast Cancer in Patients and Healthy Participants Undergoing Breast Cancer Screening, Breast Diagnostic Studies, or Treatment for Benign Breast Disease
Status: Terminated | Type: Observational
Why Stopped: Closed due to low accrual
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00080; P30CA033572 (NIH); CHNMC-00080; CDR0000629067 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-12-20; First posted 2008-12-23 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ | interventions — Immunohistochemistry; Chromatography, Liquid; Mass Spectrometry; Biopsy, Fine-Needle; Biopsy, Needle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal participants
  Interventions: Genetic: protein analysis; Genetic: protein expression analysis; Genetic: proteomic profiling; Other: diagnostic laboratory biomarker analysis; Other: immunohistochemistry staining method; Other: liquid chromatography; Other: mass spectrometry; Procedure: fine-needle aspiration; Procedure: needle biopsy; Procedure: radiomammography
- Breast Cancer Patients
  Interventions: Genetic: protein analysis; Genetic: protein expression analysis; Genetic: proteomic profiling; Other: diagnostic laboratory biomarker analysis; Other: immunohistochemistry staining method; Other: liquid chromatography; Other: mass spectrometry; Procedure: fine-needle aspiration; Procedure: needle biopsy; Procedure: radiomammography

INTERVENTIONS:
Genetic: protein analysis — protein analysis
Genetic: protein expression analysis — protein expression analysis
Genetic: proteomic profiling — proteomic profiling
Other: diagnostic laboratory biomarker analysis — Performed one time on study
Other: immunohistochemistry staining method — Performed one time on study
Other: liquid chromatography — Performed on samples collected one time on study
Other: mass spectrometry — Performed on samples collected one time on study
Procedure: fine-needle aspiration — Samples collected one time on study at the appointment for fine-needle aspiration where applicable
Procedure: needle biopsy — Samples collected one time on study at the appointment for needle biopsy where applicable
Procedure: radiomammography — Samples collected one time on study at the appointment for radiomammography where applicable

SUMMARY:
RATIONALE: Diagnostic procedures that measure biomarker levels in nipple section and blood samples, may help in the early detection of breast cancer.

PURPOSE: This clinical trial is studying nipple secretion samples in detecting breast cancer in patients and healthy participants undergoing breast cancer screening, breast diagnostic studies, or treatment for benign breast disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine CEA levels in nipple secretions and blood samples from breast cancer patients and normal controls.
* To determine the sensitivity and specificity of measuring CEA levels in nipple secretions and blood samples for the detection of breast cancer.
* To validate the optical biosensor CEA levels measured in blood and nipple secretions in breast cancer patients and normal controls compared with standard protein assays.
* To develop a profile of proteins present in affected vs unaffected breasts using mass spectrometry.

OUTLINE: Patients and participants undergo nipple secretion and blood sample collection at baseline and at 1 month for evaluation of levels of carcinoembryonic antigen (CEA) and patterns of protein expression that may indicate the presence of early-stage breast cancer. Nipple secretions are obtained from both the affected and unaffected breasts via capillary, aspiration (nipple aspirate fluid [NAF]), and nipple blot . CEA levels are measured in serum samples, NAF, and other nipple secretions using standard CEA protein assays. Nipple secretions obtained by nipple blot are analyzed by nipple blot assay to determine the feasibility of using this technique. The results of the nipple blot assay are then compared with the results of standard protein assays to evaluate the sensitivity and specificity of the nipple blot test. CEA expression is also determined in breast tissue specimens obtained from patients undergoing diagnostic biopsy. Specimens are examined by IHC for tissue CEA levels. Proteomic profiles in NAF and serum samples are measured using liquid chromatography mass spectrometry and then compared with proteomic profiles in normal healthy controls.

Once the feasibility of the nipple blot assay has been determined, an optical biosensor will be developed to detect fluorescent-labeled antibodies directed against CEA found in serum and breast sections. Optical biosensor CEA levels measured in breast cancer patients and normal controls will then be compared to standard protein assays for evaluation of the sensitivity and specificity of biosensor measurements.

After completion of study intervention, patients and participants are followed for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Referred to the Women's Health Center at the City of Hope National Medical Center for breast cancer screening, breast diagnostic studies, or treatment of breast disease
* Meets 1 of the following criteria:

  * Asymptomatic and undergoing screening mammography (normal controls)
  * Symptomatic and undergoing diagnostic mammography
  * History of an abnormal mammogram and undergoing stereotactic or ultrasound-guided fine-needle aspiration or core needle biopsy
  * Recently diagnosed biopsy-proven unilateral breast cancer prior to initiation of surgical or systemic therapy
* No prior breast surgery or surgical biopsy that removed the current breast pathology
* No prior breast reconstruction or breast reduction surgery that altered the ductal drainage pattern in the affected breast

PATIENT CHARACTERISTICS:

* No other cancer within the past 5 years except skin cancer
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2001-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
CEA levels in nipple secretions and blood samples from breast cancer patients and normal controls | Baseline
Sensitivity and specificity of measuring CEA levels in nipple secretions and blood samples from breast cancer patients and normal controls | Baseline
Comparison of optical biosensor CEA levels with CEA levels measured by standard protein assays in blood samples and nipple secretions from breast cancer patients and normal controls | Baseline
Profile of proteins present in fluid from affected vs unaffected breasts as assessed by mass spectrometry | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: John Yim, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States